CLINICAL TRIAL: NCT03947541
Title: Utility of Postoperative Bracing: A Single-institution, Randomized-control Trial Comparing Brace to No-brace for Patients Undergoing Long-segment Fusion for Spinal Deformity
Brief Title: Utility of Postoperative Bracing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00100497
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Bracing for Spinal Deformity
Keywords: Thoracolumbosacral (TLSO) brace; Lumbosacral orthotic (LSO) brace; Adult spinal deformity; Postoperative Brace
MeSH Terms: interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Brace (Active Comparator): Patients randomized to the no-brace group will not be required to wear a brace, postoperatively.
  Interventions: Other: No Bracing
- Brace (Experimental): Patients randomized to the brace group will wear the brace when out of bed and will be allowed to remove the brace when in bed. This intervention will continue through their 6-week postoperative visit, after which point, patients will be allowed to wear the brace for comfort.
  Interventions: Other: Thoracolumbosacral (TLSO) brace

INTERVENTIONS:
Other: Thoracolumbosacral (TLSO) brace — Patients will be required to wear the TLSO brace when out of bed, beginning on postoperative day 2 through 6 week follow-up period.
  Arms: Brace
Other: No Bracing — Participants will not wear a brace in the study.
  Arms: No Brace

SUMMARY:
The study is being done to assess if the use of bracing helps improve quality of life of patients that are undergoing a spinal fusion for deformity.

If the participant agrees to be in this trial they will be randomly assigned (like the flip of a coin) to receive either brace treatment or non-brace treatment.

Regardless of what treatment group the participants are in, they will undergo surgery as planned. After surgery, patients in both groups will be treated per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* The principal investigator's new or returning patients
* Adults 18 to 80 years of old
* Undergoing a spinal fusion procedure of greater than or equal to 5 levels for the purpose of correcting idiopathic spinal deformity

Exclusion Criteria:

* Patients who are undergoing a spinal fusion for other reasons besides deformity
* Patients who are unable to provide consent or fill out survey questionnaires
* Patients who have brace-prohibitive body habitus
* Patients who are unable to obtain standing AP and lateral 3-foot standing scoliosis x-rays

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) score | Baseline, 3 months, 6 months, 12 months and 24 months
  Scores from 0 to 5, and the total is added and multiplied by 2. Therefore, the ODI ranges from 0 to 100. A higher score on the ODI indicates a more severe disability.

SECONDARY OUTCOMES:
Changes in Scoliosis Research Society Outcomes Questionnaire (SRS-22 and SRS-30) | Baseline, 3 months, 6 months, 12 months and 24 months
  Measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions). The maximum score in each domain is 5 and minimum score is 1, with higher scores representing greater patient quality of life.
Change in Visual Analogue Scale (VAS) | Baseline, 3 months, 6 months, 12 months and 24 months
  Scale from 0 to 10, 0 being no pain and 10 being worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Karikari, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No